CLINICAL TRIAL: NCT06428851
Title: Comparison of Laser Therapy Versus Neuromuscular Electrical Nerve Stimulation at Hemiplegic Shoulder Pain and Upper Extremity Functions
Brief Title: Laser Therapy Versus Neuromuscular Electrical Nerve Stimulation at Hemiplegic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Pınar Özge Başaran, Principal Investigator, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-174
Record Dates: First submitted 2024-05-17; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Hemiplegic Shoulder Pain
Keywords: hemiplegic shoulder pain; electrical nerve stimulation; laser
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: 1. Laser therapy
  2. Neuromuscular electrical nerve stimulation therapy (NMES)
  3. Control: classical physical therapy exercises
  3)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants: stroke patients with shoulder pain Care provider: physiotherapist who applied the treatments to the patients Investigator: Researchers who were blinded to the treatment groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser therapy Group (Active Comparator): Classical physical therapy exercises were applied according to the patient's needs and neurologic level. These exercises are determined by the physiotherapist according to the functional status of the patient and consist of passive, passive assisted, active range of motion exercises, stretching and strengthening exercises, mobilization exercises. Group 1 Laser therapy group (n:25) in addition to classical physical therapy, laser was applied to the shoulder group muscles for 5 minutes a day, 3 days a week for 4 weeks.
  Interventions: Other: Laser therapy
- Neuromuscular electrical nerve stimulation Group (Active Comparator): Classical physical therapy exercises were applied according to the patient's needs and neurologic level. These exercises are determined by the physiotherapist according to the functional status of the patient and consist of passive, passive assisted, active range of motion exercises, stretching and strengthening exercises, mobilization exercises. In Neuromuscular electrical nerve stimulation group, in addition to these exercises, Neuromuscular electrical nerve stimulation was applied to the shoulder flexor and abductor muscle groups for 20 minutes a day, 5 days a week for a total of 4 weeks.
  Interventions: Other: Neuromuscular electrical nerve stimulation
- Control Group (Active Comparator): Classical physical therapy exercises were applied according to the patient's needs and neurologic level. These exercises are determined by the physiotherapist according to the functional status of the patient and consist of passive, passive assisted, active range of motion exercises, stretching and strengthening exercises, mobilization exercises.
  Interventions: Other: Control

INTERVENTIONS:
Other: Laser therapy — Shoulder girdle muscles were lasered for 5 minutes a day, 3 days a week, total of 4 weeks.
  Arms: Laser therapy Group
Other: Neuromuscular electrical nerve stimulation — Neuromuscular electrical nerve stimulation was applied to the shoulder flexor and abductor muscles for 20 minutes a day 5 days a week, total of 4 weeks.
  Arms: Neuromuscular electrical nerve stimulation Group
Other: Control — Classical physical therapy exercises were applied according to the patient's needs and neurologic level. These exercises are determined by the physiotherapist according to the functional status of the patient and consist of passive, passive assisted, active range of motion exercises, stretching and strengthening exercises, mobilization exercises 5 days a week for 1 hour, total of 4 weeks.
  Arms: Control Group

SUMMARY:
This study aimed to investigate whether laser and neuromuscular electrical nerve stimulation applied in addition to conventional physical therapy exercises in hemiplegic shoulder pain seen in patients with stroke provides an additional contribution to pain, range of motion, spasticity, upper extremity functions and whether the two treatment types are superior to each other.

DETAILED DESCRIPTION:
Cerebrovascular events, which are estimated to affect approximately 9 million people worldwide, have emerged as a serious cause of morbidity and mortality due to prolonged human lifespan. With the use of effective treatment methods in acute treatment, the level of expectation regarding prognosis has increased. Secondary complications that develop after stroke are frequently encountered. These complications cause serious disruptions in the rehabilitation process. The upper extremity is affected more frequently than the lower extremity and recovery is more difficult and slower. Most of the functional impairments related to the upper extremity are shoulder problems. The most important reason is impaired shoulder biomechanics. Pain may occur in the first 2 weeks after stroke or typically occurs 1 to 3 months after stroke. Pain in the hemiplegic shoulder significantly reduces patients' function and rehabilitation capacity. Reducing pain with effective methods applied for pain increases participation in rehabilitation and increases the range of motion measurements and functional capacity.

There are many physical therapy approaches in the treatment of hemiplegic shoulder pain. Light amplification by stimulated emission of radiation (laser) is one of these treatment approaches and briefly means intensified light. Laser principles are based on the quantum concept introduced by Einstein in 1927. Theodore Maiman developed the first laser device in 1960. According to the basic working principle of laser devices; the photon energy emitted from a light source is passed through a specific medium and it is thought to be effective in reducing pain in the tissue, increasing the range of motion, and improving upper extremity functions. As a result of all these mechanisms of action, laser beams are used in medicine to utilize their regenerative, biostimulating, analgesic, anti-inflammatory, and anti-edematous effects. These laser methods have been previously studied in knee osteoarthritis and shoulder adhesive capsulitis. Laser has also been investigated in hemiplegia.

Neuromuscular electrical nerve stimulation (NMES) produces muscle contractions using electrical pulses. These electrical pulses are delivered to the current muscles through superficial electrodes. The action potential from the central nervous system is mimicked with NMES and contraction is produced in the muscle.

There is no study in the literature comparing laser and neuromuscular electrical nerve stimulation in the hemiplegic shoulder.

This study aimed to investigate whether laser and neuromuscular electrical nerve stimulation applied in addition to conventional physical therapy exercises in hemiplegic shoulder pain seen in patients with stroke provides an additional contribution to pain, range of motion, spasticity, upper extremity functions and whether the two treatment types are superior to each other. In this prospective randomized controlled study, 75 stroke patients aged 18-85 years with shoulder pain who were diagnosed with ischemic stroke for the first time and who applied to the Physical Therapy and Rehabilitation Outpatient Clinic between December 2023 and May 2024 were included in the study. The patients included in the study were divided into 3 groups by the same physiotherapist by envelope drawing method. Due to the nature of the study, the physiotherapist administering the treatment was aware of the groups of the patients. On the other hand, all evaluations were performed by the same researcher who was blinded to the type of treatment. All patients underwent a multidisciplinary rehabilitation program 5 days a week for 4 weeks for a total of 20 sessions. Classical physical therapy exercises were applied according to the patient's needs and neurologic level. These exercises are determined by the physiotherapist according to the functional status of the patient and consist of passive, passive assisted, active range of motion exercises, stretching and strengthening exercises, mobilization exercises. 1st group laser group (n:25) received laser for 5 minutes a day 3 days a week in addition to classical physical therapy, 2nd group ES group (n:25) received Neuromuscular electrical nerve stimulation for 20 minutes a day 5 days a week in addition to classical physical therapy. 3. Group, control group (n:25), classical physical therapy exercises were applied.

ELIGIBILITY:
Inclusion Criteria

* diagnosed with unilateral ischemic stroke for the first time
* 18-85 years old,
* patients with shoulder pain

Exclusion Criteria:

* another disease that will affect the central nervous system
* injections or physical therapy to the same shoulder in the last 3 months,
* history of shoulder surgery,
* cervical radiculopathy,
* inflammatory rheumatic disease or infection,
* serious cardiovascular disease such as heart failure, arrhythmia, myocardial infarction that will affect functional status,
* disease that will cause cognitive dysfunction,
* Alzheimer's disease, dementia,
* severe visual loss,
* pregnancy and lactation,
* malignancy,
* psychiatric diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Pain Level | baseline and through study completion, an average of 4 weeks
  The pain level of the patients will be measured with a scale given to the patient; visual pain scale. Patients rate their pain on a scale of 0-10. It consists of scores ranging from 0 (no pain) to 10 (most severe pain). Higher scores indicate more severe pain.

SECONDARY OUTCOMES:
upper extremity functions | baseline and through study completion, an average of 4 weeks
  upper extremity functions were evaluated with Fugl-Meyer. Fugl-Meyer is a stroke-specific performance-based scale, fully filled by the same investigator, each parameter is scored between 0-2. The total score is between 0 to 100. 0: unsuccessful, 1: partially successful, 2: completely successful performance. A higher score indicates better performance
Disability | baseline and through study completion, an average of 4 weeks
  he Shoulder Pain and Disability Index is a patient-completed scale consisting of 5 items on pain and 8 items on disability. Each item is marked by the patient on a 0-10 cm scale. High scores indicate high pain and disability.
Daily living activities | baseline and through study completion, an average of 4 weeks
  Barthel index It is filled out after the examination by the same investigator to evaluate the activities of daily living of the patients. Turkish version of the scale has been adapted. The Barthel index consists of 10 items related to activities of daily living and mobility. Nutrition, transition from wheelchair to bed and back, self-care, bathing, walking, climbing up and down stairs, dressing, bladder and bowel continence are evaluated. The items can be divided into two parts related to self-care and mobility. A scoring is based on whether the person is assisted in performing these tasks. The highest total score that can be achieved is 100, which means that the individual is completely independent in their physical functioning. The lowest score is 0, indicating that the individual is completely dependent
Spasticity | baseline and through study completion, an average of 4 weeks
  The Modified Ashworth Scale, the most widely used scale for tonus assessment, was used to evaluate spasticity. In this scale, muscle tone is evaluated between 0 normal and 4 being rigid. In our study, spasticity in shoulder adductors and internal rotators, forearm flexors, wrist flexors and finger flexors were recorded by the same investigator.
Recovery Stage | baseline and through study completion, an average of 4 weeks
  Brunnstrom Recovery Stage is a 6-step scale that includes movement patterns with progressively increasing recovery evaluated separately for upper extremity, hand and lower extremity. 0: no movement, 6: full movement. Higher values indicate better motor recovery and were recorded by the same investigator.

CONTACTS AND LOCATIONS:
Overall Officials: MUSTAFA KESER, Ass Prof, Study Chair — HİTİT UNİVERSİTY EROL OLÇOK RESEARCH HOSPİTAL
Locations (1):
- Hitit University, Çorum, Turkey (Türkiye)